CLINICAL TRIAL: NCT02860793
Title: Role of PTK-7 in Acute Myeloid Leukemias: Impact of PTK7 Serum Marker and ex Vivo Studies to Decipher the Role of PTK7
Brief Title: Role of PTK-7 in Acute Myeloid Leukemias
Acronym: LAM-PTK7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LAM-PTK7-IPC 2013-011
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: PTK7; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AML patients at diagnosis (Experimental)
  Interventions: Other: Bone marrow aspiration; Other: Blood sampling

INTERVENTIONS:
Other: Bone marrow aspiration
Other: Blood sampling

SUMMARY:
The pseudo tyrosine kinase receptor 7 (PTK7) is an orphan tyrosine kinase receptor assigned to the planar cell polarity pathway. PTK7 is expressed in normal myeloid progenitors and CD34(+) CD38(-) bone marrow cells in humans. It is also expressed in acute myeloid leukemia (AML) and is mostly assigned to granulocytic lineage differentiation. In AML, PTK7 seems to convey promigratory and antiapoptotic signals into the cell and represents an independent prognosis factor of survival in patients treated with induction chemotherapy. This study aims at:

* evaluating the impact of PTK7 expression on primary AML cells ex vivo
* evaluating the diagnostic and prognostic value of a soluble form of PTK7

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* AML at diagnosis, not previously treated
* Treatment by induction chemotherapy
* Signed informed consent
* Affiliation to the French social security system

Exclusion Criteria:

* pregnant woman(or of childbearing potential) or breastfeeding woman
* emergency
* patients deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Evaluation PTK7+ and PTK7- AML cells hematopoietic homing abilities in xenografted mice by in vivo bioluminescence imaging | 1 day
Soluble PTK7 measurement in the serum | 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Norbert VEY, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches du Rhone, France

IPD SHARING:
Plan to Share IPD: No